CLINICAL TRIAL: NCT03689075
Title: Study to Compare Once-daily Extended Release Tacrolimus Versus Twice-daily Immediate Release Tacrolimus Following Renal Allograft Failure to Reduce the Risk of Allosensitisation
Brief Title: Extended Release Versus Immediate Release Tacrolimus Following Renal Allograft Failure to Reduce Allosensitisation
Acronym: EVITRA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Non-feasible due to change in clinical practice
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18IC4423
Record Dates: First submitted 2018-09-20; First posted 2018-09-28 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Kidney Transplant Failure; Allosensitization; Immunosuppression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate release tacrolimus (No Intervention): Patients will continue on immediate release tacrolimus
- Extended release tacrolimus (Active Comparator)
  Interventions: Drug: Envarsus Oral Product

INTERVENTIONS:
Drug: Envarsus Oral Product — Patients will be randomised to receive either envarsus or to continue on an immediate release tacrolimus formulation
  Arms: Extended release tacrolimus

SUMMARY:
Study to compare once-daily extended release tacrolimus versus twice-daily immediate release tacrolimus following renal allograft failure to reduce the risk of allosensitisation

ELIGIBILITY:
Inclusion Criteria:

1. Able to give informed consent.
2. Male or female, at least 18 years of age.
3. Has renal allograft failure and is due to start haemodialysis therapy or within 28 days following starting dialysis.
4. Has been already activated on the transplant wait list or is undergoing work up to be reactivated on the transplant list.
5. Has no indication for graft nephrectomy at the time of transplant failure.
6. Is receiving an immediate release tacrolimus maintenance immunotherapy regimen at the time of allograft failure.

Exclusion Criteria:

1. Has another functioning organ transplanted (eg. pancreas, liver, cardiac) at the time of kidney allograft failure.
2. Allograft failure within a month of transplant.
3. Patients who are due to receive or receiving peritoneal dialysis following graft failure.
4. Patients with detectable DSA at the time of allograft failure
5. Receiving an extended release preparation of tacrolimus as immunotherapy at the time of graft failure.
6. Requires continuation of maintenance immunosuppression other than prednisolone or tacrolimus (eg. Mycophenolate mofetil or sirolimus).
7. Patients who on IR-FK conversion would require less than 0.75mg of Envarsus.
8. HLA type of donor is unknown.
9. Has a history of, or active co-morbidity that in the Investigator's opinion, could affect the conduct of the study.
10. Has any condition at the time of recruitment which would prohibit or pose a relative contraindication for the continued use of tacrolimus to a target trough level of between 3-5ng/ml
11. Active bacterial, viral (including CMV and EBV) or parasitic infections, including tuberculosis that, in the Investigator's opinion, could affect the conduct of the study.
12. Has active malignancy.
13. Female patients of child bearing age, who wish to consider pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Incidence of de novo allosensitisation (donor specific antibodies) at 24 months post allograft failure. | 24 months
  Number of patients who develop new DSA in each group

SECONDARY OUTCOMES:
Medication adherence measurement | 24 months
  Will be measured by BAASIS questionnaire (comparison of scores)
Health-Related Quality of Life measurement | 24 months
  Will be measured by the EQ-5D-5L Questionnaire (comparison of scores) - 5D
  - 5L Questionnaire
Coefficient of variation of tacrolimus levels at 24 months post allograft failure. | 24 months
  Incorporating all study visit trough tacrolimus levels (standard deviation/mean)
Adverse events | 24 months
  Incidence of infective episodes, malignancy, diabetes, erythropoietin resistance, graft nephrectomy
Chances of re-transplantation as determined by the transplant matchability calculator available from NHSBT | 24 months
  Will be calculated by using the NHSBT calculator
Proportion of patients retransplanted during the study period | 24 months
  Proportion of patients in each arm receiving a transplant

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No